CLINICAL TRIAL: NCT00777348
Title: Clinical Trial to Assess the Protective Effect of the Fixed Drug Combination of Disodium Cromoglycate Plus Reproterol in Comparison to the Single Components and Placebo in Adults With Exercise Induced Asthma Randomised, Placebo-controlled, Double-blind, Crossover, Multicentre Study
Brief Title: To Assess the Protective Effect of the Fixed Drug Combination of Disodium Cromoglycate Plus Reproterol
Acronym: AERIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Collaborators: ClinResearch, GmbH (Other); Sanofi (Industry)
Responsible Party: Meda Pharma GmbH & Co. KG, Dr. DT Nguyen, Senior Medical Manager, Meda Pharma GmbH & Co. KG, Bad Homburg, Germany
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-00982-3256; EudraCT No.: 2007-002553-23
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2009-04

CONDITIONS: Asthma, Exercise-Induced
MeSH Terms: conditions — Asthma, Exercise-Induced | interventions — reproterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): DSCG + Reproterol
  Interventions: Drug: Combination DSCG and Reproterol
- 2 (Active Comparator): DSCG
  Interventions: Drug: Combination DSCG and Reproterol
- 3 (Active Comparator): Reproterol
  Interventions: Drug: Combination DSCG and Reproterol
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Combination DSCG and Reproterol

INTERVENTIONS:
Drug: Combination DSCG and Reproterol — 1:

SUMMARY:
This is a multicentre, randomised, double-blind, placebo-controlled, 4-way cross-over study. At each study visit a standardised treadmill test will be performed to provoke EIA. Before and after the challenge test pulmonary function variables (e.g. forced expiratory volume in one second (FEV1)) will be measured in order to assess the protective effect of the study medication.

DETAILED DESCRIPTION:
* Primary objective: to demonstrate superiority of the protective effect of the fixed combination of disodium cromoglycate (DSCG) plus reproterol in comparison to the single component reproterol in adults suffering from exercise induced asthma (EIA).
* Secondary objectives: to demonstrate superiority of the protective effect of DSCG plus reproterol in comparison to the single component DSCG; to demonstrate superiority of the protective effect of each single component in comparison to placebo. In addition, the tolerability of medications will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects aged 18 - 65 years
* Exercise induced asthma with reversible airway obstruction: twice proven EIA defined as maximum decrease in FEV1 against the baseline value of at least 20% (first test results can be obtained during the last 12 months)
* Baseline FEV1 before challenge must be > or = 70% of the predicted FEV1

Exclusion Criteria:

Safety concerns:

* Subjects with hypersensitivity to DSCG, reproterol, menthol, peppermint or other excipients of the study medication
* Pregnancy, breast-feeding or planned pregnancy during the study. Women of child bearing potential not using a highly effective method of birth control defined as those which result in a low failure rate (i.e. <1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, hormonal IUDs, tubal ligation or vasectomised partner
* Subjects with an asthma exacerbation within 4 weeks prior to the study start. Asthma exacerbation defined as use of oral (systemic) glucocorticosteroids, unscheduled consultation of a medic due to asthma, hospitalisation, or additional treatment of asthma with antibiotics
* Eosinophilic pneumonia
* Clinically significant cardiovascular diseases (e.g. cardiac infarction, cardiac dysrhythmia, hypertrophic obstructive cardiomyopathy, coronary heart disease…)
* Resting blood pressure over 140/90 mmHg
* Diastolic blood pressure after treadmill-test over 120 mmHg
* Malignancies including phaeochromocytoma within the last 5 years
* Severe hyperthyreosis, thyreotoxicosis, instable diabetes mellitus

Lack of suitability for the trial:

* Subjects with seasonal asthma during their asthma season
* Infectious disease of the upper airways within 2 weeks prior to the study and within 4 weeks prior to study in case of use of antibiotics
* Relevant respiratory disorder other than asthma
* Clinically significant renal, endocrine, haematological, hepatic, immunological, gastrointestinal, neurological, or psychiatric diseases
* Any chronic disease which might influence absorption, metabolism, or excretion of the trial substances
* Change of inhalative glucocorticosteroid dosage and / or antiasthmatic controller therapy within the last 4 weeks prior to or during the study
* Concomitant systemic treatment with glucocorticosteroids
* Concomitant treatment with any ß-antagonistic drug
* Need of rescue medication within 15 min after challenge
* Concomitant therapy with antidepressants or neuroleptics
* Drug or alcohol abuse which would interfere with the subjects proper completion of the protocol assignment and mentally handicapped subjects
* Smokers within the last 6 months or smoking history > 10 pack-years (a pack-year is 20 cigarettes per day for one year or equivalent)
* Exposure to another investigational agent within the last 4 weeks prior to this one or during this study
* Non-cooperative subjects not able to understand the instructions for use of the devices

Administrative reasons:

* Lack of ability or willingness to give informed consent
* Lack of willingness to have personal study related data collected, archived or transmitted according to protocol
* Anticipated non-availability for study visits / procedures
* Personnel involved in the planning or conduct of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Primary objective: to demonstrate superiority of the protective effect of the fixed combination of disodium cromoglycate (DSCG) plus reproterol in comparison to the single component reproterol in adults suffering from exercise induced asthma (EIA). | 5, 10, 15, 30 and 60 minutes after drug application

SECONDARY OUTCOMES:
Secondary objectives: to demonstrate superiority of the protective effect of DSCG plus reproterol in comparison to the single component DSCG; to demonstrate superiority of the protective effect of each single component in comparison to placebo. | 5, 10, 15, 30 and 60 minutes after drug application

CONTACTS AND LOCATIONS:
Overall Officials: Roland Buhl, MD, Prof., Principal Investigator — Clinical Research Pneumology, III. Medical Clinic, University Clinic Mainz
Locations (7):
- Germany (7):
  - Kurmittelhaus der Moderne, Bad Reichenhall
  - Asthma Center Buchenhoehe, Berchtesgaden
  - Practice Dr. T. Ginko, Bonn
  - Clinic St. Georg Leipzig, Robert Koch Clinic, Leipzig
  - Clinical Research Pneumology, III. Medical Clinic, University Clinic Mainz, Mainz
  - Practice Dr. W. Schürmann, Marburg
  - Institute for Pulmonary Research GmbH, Wiesbaden